CLINICAL TRIAL: NCT07057414
Title: Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Single-Center Clinical Study to Evaluate the Safety and Efficacy of GMDTC for Injection in Subjects With Elevated Cadmium Levels
Brief Title: The Safety and Efficacy of GMDTC for Injection in Subjects With Elevated Cadmium Levels
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Jianersheng Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: Guangdong Provincial Hospital for Occupational Disease Prevention and Treatment (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GuangdongPharm IIa
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cadmium Exceeds the Standard
Keywords: Cadmium; Cadmium Poisoning; Therapeutics; Drugs, Investigational; GMDTC
MeSH Terms: conditions — Cadmium Poisoning | interventions — Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study anticipates 11 subjects per dose group (including 3 placebo controls), with the total sample size to be determined based on actual study progress.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMDTC Group (Experimental): Participants randomized to the GMDTC Group will receive daily administrations (GMDTC for Injection ) after breakfast from Day 1 to Day 5 and Day 8 to Day 12.
  Interventions: Drug: GMDTC for injection
- Placebo Group (Placebo Comparator): Participants randomized to the Placebo Group will receive daily administrations (normal saline for Injection ) after breakfast from Day 1 to Day 5 and Day 8 to Day 12.
  Interventions: Other: 0.9% Sodium Chloride Injection(0.9% NaCl)

INTERVENTIONS:
Drug: GMDTC for injection — GMDTC for Injection with a specification of 0.5g/vial, and administered by intravenous infusion. According to the drug preparation SOP , Using 0.9% physiological saline to achieve the required concentration for each dose group (e.g., The initial dose group: 2 g reconstituted in 500 mL, with each 1 g reconstituted in 250 mL, resulting in a 4 mg/mL concentration.). All infusion-related reactions must be documented. Drug preparation must be performed by an non-blind investigator independent of the study to maintain blinding integrity for other study personnel.
  Arms: GMDTC Group
Other: 0.9% Sodium Chloride Injection(0.9% NaCl) — 0.9% Sodium Chloride Injection with a specification of 250mL/bag, and administered by intravenous infusion. The infusion should be strictly adhering to the assigned dosage. All infusion-related reactions must be documented. Drug preparation must be performed by an non-blind investigator independent of the study to maintain blinding integrity for other study personnel.
  Arms: Placebo Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-center Phase IIa clinical study.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the pharmacodynamic characteristics of GMDTC for Injection in subjects with elevated cadmium levels after administration, while the secondary objectives are to assess the safety, tolerability and pharmacokinetic profile of GMDTC for Injection following multiple-dose administration in the same population; based on the results from Phase I single- and multiple-dose studies, the initial dose group in this trial is set at 2000 mg with a concentration of 4 mg/mL, where the first 4 participants (including 3 in the treatment group and 1 in the placebo group) will be enrolled first, and subsequent participants in the same dose group can only continue enrollment after investigators complete the 72-hour post-dose safety and tolerability assessments and confirm favorable results, with the SMC meeting to determine subsequent study plans including but not limited to dose escalation, concentration adjustment or increased treatment duration after completion of observation for each dose group.

ELIGIBILITY:
Inclusion Criteria:

Study participants must meet all of the following criteria to be enrolled in this trial:

1. Voluntarily sign the informed consent form, aged between 18 and 70 years (inclusive), regardless of gender;
2. Single morning urine cadmium >5 μg/g creatinine (with creatinine concentration ≥0.3 g/L and ≤3 g/L);
3. eGFR ≥30 mL/min/1.73 m² (calculated using the CKD-EPI formula).

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Currently suffering from any clinically significant disease that, in the investigator's judgment, poses a safety risk for participation in this clinical trial;
2. Patients with a history of kidney disease requiring hemodialysis;
3. Patients with a history of severe infusion-related allergic reactions, known allergies to three or more substances, or known hypersensitivity to any component of this product (e.g., disodium edetate, mannitol);
4. Previous diagnosis of diabetes with poorly controlled blood glucose;
5. History of conditions predisposing to hypokalemia (e.g., periodic hypokalemia, primary aldosteronism);
6. High-risk uncontrolled arrhythmia within the past 6 months, including:

1) Resting atrial tachycardia with heart rate >100 bpm, 2) Significant ventricular arrhythmia (e.g., ventricular tachycardia), 3) High-grade atrioventricular block (e.g., Mobitz type II second-degree or third-degree AV block), 4) NYHA Class IV heart failure, 5) Left ventricular ejection fraction (LVEF) <50%; 7.Prolonged QT/QTc interval at screening/baseline (QTc: >450 ms in males, >470 ms in females) or known family history of long QT syndrome; 8. Use of any medication or supplement (e.g., SGLT2 inhibitors like dapagliflozin, canagliflozin, empagliflozin, etc.; GLUT2 inhibitors like cytochalasin B, phloretin, etc.) within 14 days prior to screening that may interact with the investigational drug; 9. Participation in any other clinical trial involving investigational drugs or medical devices within 3 months prior to screening; 10. Major surgery within 4 weeks before screening or planned surgery during the trial that may affect drug metabolism or safety assessment; 11. Blood donation or significant blood loss (≥200 mL, excluding menstrual bleeding), transfusion, or use of blood products within 1 month prior to screening; 12. Intolerance to venipuncture and/or history of syncope due to blood or needle exposure; 13. Pregnant or lactating women, or participants unwilling to use effective non-pharmacological contraception during the trial; 14. Inability to use contraception for 6 months after trial completion; 15.Inability to comply with dietary restrictions or nutritional guidelines; 16.Alcohol abuse or regular alcohol consumption (>14 units/week; 1 unit ≈ 200 mL beer [5%], 25 mL spirits [40%], or 85 mL wine [12%]) within 6 months before screening, or unwillingness to abstain from alcohol during the trial; 17. Participants with unstable psychiatric disorders, in the investigator's opinion, who cannot cooperate with the study; 18. Any other condition deemed by the investigator to compromise study compliance or safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic Parameters , 24-hour urinary cadmium | Evaluated at pre-dose (Day-1) and post-dose (Day1-Day6, Day8-Day13)
  24-hour urinary cadmium excretion before and after drug administration(μg/L)

SECONDARY OUTCOMES:
Adverse Events (AEs) | Within 30 days after the last dose administration
  Clinical safety assessments during the trial will include: 1) all spontaneously reported and directly observed adverse events (AEs) and serious adverse events (SAEs); 2) any clinically significant changes in vital signs (as determined by the investigator); 3) clinically significant abnormalities (as determined by the investigator) observed during physical examinations, laboratory tests, electrocardiograms (ECG), cardiac ultrasound, abdominal ultrasound, thyroid ultrasound, chest CT scans, ophthalmologic examinations, auditory tests, and olfactory tests, with AE severity graded according to CTCAE v5.0 standards.
Pharmacodynamic Parameters , Urinary Cadmium and Lead Levels | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13, Day15)
  urinary Cadmium and Lead Levels before and after drug administration (μg/g Creatinine)
Pharmacodynamic Parameters , 24-Hour Urinary Lead and Copper | Evaluated at pre-dose (Day-1) and post-dose (Day1-Day6, Day8-Day13)
  24-Hour Urinary Lead and Copper Excretion before and after drug administration(μg/L)
Pharmacodynamic Parameters , Blood Heavy Metal/Metalloid Levels(Pb, As, Hg, Cr, Mn) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13)
  Blood Heavy Metal/Metalloid Levels (Pb, As, Hg, Cr, Mn) before and after drug administration(μg/L)
Pharmacodynamic Parameters , Blood Heavy Metal/Metalloid Levels(Cu, Zn) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13)
  Blood Heavy Metal/Metalloid Levels (Cu, Zn) before and after drug administration(mg/L)
Pharmacodynamic Parameters , Renal Function Biomarker Levels(Creatinine-corrected urinary β2-MG, Creatinine-corrected urinary URBP) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13, Day15)
  Renal Function Biomarker Levels (Creatinine-corrected urinary β2-microglobulin, Creatinine-corrected URBP ) before and after drug administration (μg/g Creatinine)
Pharmacodynamic Parameters , Renal Function Biomarker Levels(β2-MG, URBP) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13, Day15)
  Renal Function Biomarker Levels (Urinary β2-microglobulin (β2MG), Urinary retinol-binding protein (URBP)) before and after drug administration(μg/L)
Pharmacodynamic Parameters , Renal Function Biomarker Levels(α1-MG) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13, Day15)
  Renal Function Biomarker Levels (Urinary α1-microglobulin) before and after drug administration(mg/L)
Pharmacodynamic Parameters , Renal Function Biomarker Levels(NAG) | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13, Day15)
  Renal Function Biomarker Levels (Urinary N-acetyl-β-D-glucosaminidase (NAG) ) before and after drug administration(U/L)
Pharmacodynamic Parameters, Bone Metabolism Biomarker Levels(PTH) | Evaluated at Pre-dose (Screening Period) and post-dose (Day6, Day13)
  Bone Metabolism Biomarker Levels(Parathyroid hormone (PTH)) before and after drug administration(pg/mL)
Pharmacodynamic Parameters, Bone Metabolism Biomarker Levels(25(OH)D, P1NP, CTX) | Evaluated at Pre-dose (Screening Period) and post-dose (Day6, Day13)
  Bone Metabolism Biomarker Levels(25-Hydroxyvitamin D, Serum procollagen type I N-terminal propeptide (P1NP), Serum C-terminal telopeptide of type I collagen (CTX)) before and after drug administration(ng/mL)
Pharmacodynamic Parameters, Bone Metabolism Biomarker Levels(ALP) | Evaluated at Pre-dose (Screening Period) and post-dose (Day6, Day13)
  Bone Metabolism Biomarker Levels(Serum alkaline phosphatase (ALP)) before and after drug administration(U/L)
Pharmacodynamic Parameters , urinary cadmium Levels | Evaluated from Baseline (Pre-dose Day1) to First Void Post-dose (Day1-Day5 & Day8-Day12)
  Change in Urinary Cadmium Levels before and after drug administration (μg/g Creatinine)
Pharmacodynamic Parameters , Blood Cadmium Concentration | Evaluated at pre-dose (Day1) and post-dose (Day6, Day8, Day13)
  Blood Cadmium (Cd) Concentration before and after drug administration(μg/L)
Pharmacokinetic Parameters , Tmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Time to reach peak concentration (observed value)
Pharmacokinetic Parameters , Cmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Peak concentration (observed value)
Pharmacokinetic Parameters , λz | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Apparent terminal elimination rate constant, derived from semi-log linear regression of elimination phase concentration points.
Pharmacokinetic Parameters , t1/2 | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Apparent terminal elimination half-life, calculated using the following equation: t1/2 = Ln(2) / λz

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Wang, M.Med., Principal Investigator — Guangdong Provincial Hospital for Occupational Disease Prevention and Treatment; Ming Huang, PhD, Principal Investigator — Guangdong Provincial Hospital for Occupational Disease Prevention and Treatment
Locations (1):
- Guangdong Provincial Hospital for Occupational Disease Prevention and Treatment, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang X, Zhu J, Zhong Z, Luo M, Li G, Gong Z, Zhang C, Fei F, Ruan X, Zhou J, Liu G, Li G, Olson J, Ren X. Mobilization and removing of cadmium from kidney by GMDTC utilizing renal glucose reabsorption pathway. Toxicol Appl Pharmacol. 2016 Aug 15;305:143-152. doi: 10.1016/j.taap.2016.06.001. Epub 2016 Jun 6. PMID 27282297